CLINICAL TRIAL: NCT04631809
Title: Computer tomoGRaphy guidEd invasivE Coronary Angiography in patiEnts With a Previous Coronary Artery Bypass Graft Surgery Trial
Brief Title: Computed Tomography Coronary Angiography in Patients With a Previous Coronary Artery Bypass Graft Surgery Trial
Acronym: GREECE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Grigorios Tsigkas, assistant Professor of Cardiology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24798/28-9-2020
Record Dates: First submitted 2020-11-07; First posted 2020-11-17 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Bypass Surgery
Keywords: coronary angiography; CT-Coronary Angiography; Post-artery bypass graft surgery; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- invasive Coronary Angiography alone (Active Comparator)
  Interventions: Procedure: Coronary angiography +/- percutaneous coronary intervention
- CT-Coronary Angiography + invasive Coronary Angiography (Experimental)
  Interventions: Procedure: CT-Coronary Angiography + Coronary angiography +/- percutaneous coronary intervention

INTERVENTIONS:
Procedure: Coronary angiography +/- percutaneous coronary intervention — Comparison of performing invasive Coronary Angiography alone with performing CT-Coronary Angiography prior to the invasive Coronary Angiography
  Arms: invasive Coronary Angiography alone
Procedure: CT-Coronary Angiography + Coronary angiography +/- percutaneous coronary intervention — Comparison of performing invasive Coronary Angiography alone with performing CT-Coronary Angiography prior to the invasive Coronary Angiography
  Arms: CT-Coronary Angiography + invasive Coronary Angiography

SUMMARY:
This randomized, multi-center, prospective study seeks to compare the conventional invasive Coronary Angiography with the recently described method of performing CT-Coronary Angiography prior to the invasive Coronary Angiography, in post - CABG patients subjected to coronary angiography or percutaneous coronary intervention.

DETAILED DESCRIPTION:
Conventional invasive coronary angiography is currently used to depict coronary arteries, however in recent years, the use of CT-coronary angiography has emerged in the literature for being a non-invasive and well tolerated examination, with imaging findings often equivalent to standard coronary angiography, especially for imaging grafts in patients undergone coronary artery bypass graft surgery (CABG).

These patients present with complex anatomy of the coronary arteries making invasive coronary angiography a demanding and time-consuming examination in which the patient is exposed to large doses of radiation and volume of contrast.

Multislice computed tomography shows high diagnostic accuracy in the detection of obstruction of the grafts while the advancement of technology continuously improves the diagnostic accuracy of the imaging findings. Of course, axial coronary angiography is more sensitive and specialized in the imaging of grafts, compared to the native coronary arteries of the heart.

Therefore, the use of CT-coronary angiography before performing the respective invasive procedure is believed that it may reduce the overall duration of the procedure, the radiation received by the patient and the amount of contrast administered.

The aim of the present study is to compare the performance of CT-coronary angiography before invasive coronary angiography compared with the performance of invasive coronary angiography alone. Τhe extent to which the information obtained from CT-coronary angiography contributes to the guidance of invasive coronary angiography that will follow will be studied, regarding the total procedure time, the volume of the contrast administered the radiation to which the patient is exposed and the patient's course over a period of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Prior CABG-operation
* Age>18 years
* Indication for coronary angiography
* Informed consent

Exclusion Criteria:

* STEMI
* NSTEMI very high risk or high risk (GRACE score >140, dynamic new ST/T ECG changes)
* Hemodynamic instability
* High probability of patient's non-compliance with the study's procedures.
* Severe kidney disease with GFR<30 mL/min/1.73m2
* Known allergic reaction to contrast
* Uncontrolled Arrhythmias (mostly afib) with heart rate over 80 bpm or frequent ectopic beats which could affect the ECG-gated cCTA protocol.
* BMI>40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Total volume of contrast administered | Immediately post-procedurally

SECONDARY OUTCOMES:
Number of catheters used | Immediately post-procedurally
Total Fluoroscopy time | Immediately post-procedurally
Total Radiation Dose (Effective Dose) | Immediately post-procedurally
Total Procedure time (coronary angiography and possible angioplasty) | Immediately post-procedurally
Rate of complications related to coronary angiography (aortic dissection, coronary artery dissection, stroke, bleeding, puncture site complication) | 1-6 hours
Overall diagnostic accuracy of CTCA for estimation of graft patency will be measured, using sensitivity, specificity, positive predictive value and negative predictive value. | Immediately post-procedurally
Rate of patient survival after procedure and occurrence of major adverse cardiovascular events (MACEs). (Death, hospitalization for cardiovascular reason, re-infarction, need for revascularization, stroke) | 3-5 days
Patient survival after procedure and occurrence of major adverse cardiovascular events (MACEs). (Death, hospitalization for cardiovascular reason, re-infarction, need for revascularization, stroke). | 30 days
Rate of contrast induced nephropathy defined as increase of serum Cr of 25% or more, or an absolute increase of 0.5 mg/dl or more from baseline value, at 48-72 h following the exposure to contrast medium. | 3-5 days
Total volume of contrast agent administered during coronary angiography | Immediately post-procedurally
Total Radiation Dose (Effective Dose) during coronary angiography | Immediately post-procedurally
Number of catheters used during coronary angiography | Immediately post-procedurally

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Tsigkas, MD, PhD, Principal Investigator — University Hospital of Patras; Periklis Davlouros, MD, PhD, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yang FB, Guo WL, Sheng M, Sun L, Ding YY, Xu QQ, Xu MG, Lv HT. Diagnostic accuracy of coronary angiography using 64-slice computed tomography in coronary artery disease. Saudi Med J. 2015 Oct;36(10):1156-62. doi: 10.15537/smj.2015.10.12415. PMID 26446324
- [Background] Gaudio C, Pelliccia F, Evangelista A, Tanzilli G, Paravati V, Pannarale G, Pannitteri G, Barilla F, Greco C, Franzoni F, Speziale G, Pasceri V. 320-row computed tomography coronary angiography vs. conventional coronary angiography in patients with suspected coronary artery disease: a systematic review and meta-analysis. Int J Cardiol. 2013 Sep 30;168(2):1562-4. doi: 10.1016/j.ijcard.2012.12.067. Epub 2013 Jan 22. No abstract available. PMID 23347611
- [Background] Delewi R, Hoebers LP, Ramunddal T, Henriques JP, Angeras O, Stewart J, Robertsson L, Wahlin M, Petursson P, Piek JJ, Albertsson P, Matejka G, Omerovic E. Clinical and procedural characteristics associated with higher radiation exposure during percutaneous coronary interventions and coronary angiography. Circ Cardiovasc Interv. 2013 Oct 1;6(5):501-6. doi: 10.1161/CIRCINTERVENTIONS.113.000220. Epub 2013 Sep 24. PMID 24065442
- [Background] Dikkers R, Willems TP, Tio RA, Anthonio RL, Zijlstra F, Oudkerk M. The benefit of 64-MDCT prior to invasive coronary angiography in symptomatic post-CABG patients. Int J Cardiovasc Imaging. 2007 Jun;23(3):369-77. doi: 10.1007/s10554-006-9170-z. Epub 2006 Nov 4. PMID 17086363
- [Background] Chazen JL, Prince MR, Yip R, Min JK, Weinsaft JW, Henschke CI, Cham MD. Post-CABG coronary CT angiography: radiation dose and graft image quality in retrospective versus prospective ECG gating. Acad Radiol. 2010 Sep;17(9):1122-7. doi: 10.1016/j.acra.2010.04.011. Epub 2010 Jun 12. PMID 20542451
- [Background] Lee R, Lim J, Kaw G, Wan G, Ng K, Ho KT. Comprehensive noninvasive evaluation of bypass grafts and native coronary arteries in patients after coronary bypass surgery: accuracy of 64-slice multidetector computed tomography compared to invasive coronary angiography. J Cardiovasc Med (Hagerstown). 2010 Feb;11(2):81-90. doi: 10.2459/JCM.0b013e32832f3e2e. PMID 19851118
- [Background] Jones DA, Castle EV, Beirne AM, Rathod KS, Treibel TA, Guttmann OP, Moon JC, Smith EJ, Bourantas CV, Davies LC, Wragg A, Pugliese F, Mathur A. Computed tomography cardiac angiography for planning invasive angiographic procedures in patients with previous coronary artery bypass grafting. EuroIntervention. 2020 Feb 7;15(15):e1351-e1357. doi: 10.4244/EIJ-D-18-01185. PMID 31235457
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Tsigkas G, Makris A, Tsiafoutis I, Koutouzis M, Hamilos M, Katsanos K, Ziakas A, Brilakis ES, Davlouros P, Hahalis G. The L-RECORD Study. JACC Cardiovasc Interv. 2020 Apr 27;13(8):1014-1016. doi: 10.1016/j.jcin.2020.02.013. No abstract available. PMID 32327086
- [Background] Michael TT, Alomar M, Papayannis A, Mogabgab O, Patel VG, Rangan BV, Luna M, Hastings JL, Grodin J, Abdullah S, Banerjee S, Brilakis ES. A randomized comparison of the transradial and transfemoral approaches for coronary artery bypass graft angiography and intervention: the RADIAL-CABG Trial (RADIAL Versus Femoral Access for Coronary Artery Bypass Graft Angiography and Intervention). JACC Cardiovasc Interv. 2013 Nov;6(11):1138-44. doi: 10.1016/j.jcin.2013.08.004. Epub 2013 Oct 16. PMID 24139930
- [Background] Trattner S, Halliburton S, Thompson CM, Xu Y, Chelliah A, Jambawalikar SR, Peng B, Peters MR, Jacobs JE, Ghesani M, Jang JJ, Al-Khalidi H, Einstein AJ. Cardiac-Specific Conversion Factors to Estimate Radiation Effective Dose From Dose-Length Product in Computed Tomography. JACC Cardiovasc Imaging. 2018 Jan;11(1):64-74. doi: 10.1016/j.jcmg.2017.06.006. Epub 2017 Aug 16. PMID 28823748
- [Background] Einstein AJ, Moser KW, Thompson RC, Cerqueira MD, Henzlova MJ. Radiation dose to patients from cardiac diagnostic imaging. Circulation. 2007 Sep 11;116(11):1290-305. doi: 10.1161/CIRCULATIONAHA.107.688101. No abstract available. PMID 17846343
- [Background] Tsigkas G, Apostolos A, Synetos A, Latsios G, Toutouzas K, Xenogiannis I, Hamilos M, Sianos G, Ziakas A, Tsiafoutis I, Koutouzis M, Toulgaridis F, Moulias A, Sideris A, Patsilinakos S, Kanakakis I, Zampakis P, Tsioufis K, Kochiadakis G, Alexopoulos D, Davlouros P; GREECE Collaborators; Kalogeropoulou C, Vasilagkos G, Koufou EE, Papanikolaou A, Spanou E, Gerakaris A, Chlorogiannis D, Spiropoulou P, Miliordos I, Benetos G, Pappas C, Argentos S, Skalidis E, Kladou E, Skiadas C, Karagiannidis E, Mylona S, Zacharoulis A, Pappas L, Mantis C, Fagrezos D, Manouvelou S, Sertedaki E. Computed tomoGRaphy guidEd invasivE Coronary angiography in patiEnts with a previous coronary artery bypass graft surgery trial (GREECE trial): Rationale and design of a multicenter, randomized control trial. Hellenic J Cardiol. 2021 Nov-Dec;62(6):470-472. doi: 10.1016/j.hjc.2021.01.001. Epub 2021 Jan 20. No abstract available. PMID 33482363
- [Derived] Tsigkas G, Toulgaridis F, Apostolos A, Kalogeropoulos A, Karamasis GV, Vasilagkos G, Pappas L, Toutouzas K, Tsioufis K, Korkonikitas P, Tsiafoutis I, Hamilos M, Ziakas A, Kanakakis I, Moulias A, Zampakis P, Davlouros P. CCTA-Guided Invasive Coronary Angiography in Patients With CABG: A Multicenter, Randomized Study. Circ Cardiovasc Interv. 2024 Sep;17(9):e014045. doi: 10.1161/CIRCINTERVENTIONS.124.014045. Epub 2024 Sep 17. PMID 39286899